CLINICAL TRIAL: NCT04950491
Title: Patient-reported Outcome Measures (PROMs) Comparing Static Computer-aided Implant Surgery (s-CAIS) and Conventional Implant Surgery (CIS) for Single-tooth Replacement: A Randomized Controlled Trial
Brief Title: Patient-reported Outcome Measures Comparing Static Computer-aided Implant Surgery and Conventional Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Principal Investigator, Akarin Santivitoonvong, Doctor of Dental Surgery, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DT 071/2019
Record Dates: First submitted 2021-06-23; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Dental Implantation; Postoperative Pain; Computer-assisted Surgery; Patient Outcome Assessment; Dental Anxiety; Quality of Life; Oral Health
Keywords: Clinical Research; Dental Implant; Static Computer-Aided Implant Surgery (s-CAIS); Patient-Reported Outcome Measures (PROMs); Dental Anxiety; Pain; Oral Health-Related Quality of Life (OHRQoL)
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Surveys and Questionnaires; Quality of Life

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (s-CAIS) (Experimental): The test group workflow used a fully computer-guided implant surgical protocol.
  Interventions: Other: Modified Dental Anxiety Score (MDAS) questionnaire; Other: Pain questionnaire; Other: Oral Health-Related Quality of Life (OHRQoL) questionnaire
- Control group (CIS) (Other): The control group workflow used a conventional implant surgical protocol.
  Interventions: Other: Modified Dental Anxiety Score (MDAS) questionnaire; Other: Pain questionnaire; Other: Oral Health-Related Quality of Life (OHRQoL) questionnaire

INTERVENTIONS:
Other: Modified Dental Anxiety Score (MDAS) questionnaire — MDAS was used to measure the patients' anxiety toward dental treatment before implant surgery (Humphris, Dyer, &Robinson, 2009). Originally, the MDAS questionnaire included five questions answered with a 5-category Likert scale. The original MDAS questionnaire does not cover anxiety toward implant surgery. Therefore, a question enquiring about patients' feelings towards implant surgery was added.
Other: Pain questionnaire — Patients were asked to describe the worst pain feeling using a standard 10 cm Visual Analog Scale (VAS) and the proportion of time spent in severe pain using a 5 category Likert scale. The number of analgesics taken per day was also asked.
Other: Oral Health-Related Quality of Life (OHRQoL) questionnaire — The OHRQoL comprises 14 questions covering problems the patient may in three main categories: oral function, daily activity, and post-operative symptoms (Chaushu, Becker, Zeltser, Vasker, & Chaushu, 2004). Patients answered using a 5-category Likert scale.

SUMMARY:
The aim of this randomized controlled trial was to compare PROMs in patients receiving single tooth replacement in posterior sites by s-CAIS and CIS.

DETAILED DESCRIPTION:
Since current patient-reported outcome measures (PROMs) evidence related to static computer-aided implant surgery (s-CAIS) compared with conventional implant surgery (CIS), particularly in partial edentulous patients, were still limited. The aim of this randomized controlled trial was to compare PROMs in patients receiving single tooth replacement in posterior sites by s-CAIS and CIS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or well-controlled systemic disease (ASA classification I,II)
* A partially edentulous ridge in the premolar-molar region with existing two-sided interproximal as well as antagonist contacts
* No sign of acute oral infection
* Periodontally healthy (or successfully treated)
* More than 2 mm of keratinized gingiva at the site of surgery
* Sufficient bony ridge for implant placement with or without simultaneous bone grafting

Exclusion Criteria:

* Diabetes mellitus
* Smoking more than ten cigarettes per day
* Pregnancy
* Psychiatric disorder
* History of radiation therapy at head and neck area and chemotherapy
* Bony pathologies, namely osseous dysplasia, odontogenic cyst, tumor
* History of soft tissue grafting at the prospective implant site
* Inadequate bony ridge with the need of bone augmentation prior to implant placement

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Change of post-operative pain for 7 days: Visual Analog Scale | Patients were instructed to answer every day for 7 days starting from the day of surgery 1 hour before bedtime.
  Patients were asked to describe the worst post-operative pain feeling using a standard 10 cm Visual Analog Scale.
Change of the proportion of time spent in severe pain for 7 days: 5-category Likert scale | Patients were instructed to answer every day for 7 days starting from the day of surgery 1 hour before bedtime.
  Patients were asked to describe the proportion of time spent in severe pain using 5-category Likert scale (None, Low, Moderate, High, Very high).
Change of the analgesics taken per day for 7 days: the number of tablets per day | Patients were instructed to answer every day for 7 days starting from the day of surgery 1 hour before bedtime.
  Patients were asked to describe the number of analgesics taken per day.
Change of Oral Health-Related Quality of Life (OHRQoL) for 7 days: 5-category Likert scale | Patients were instructed to answer the OHRQoL every day for 7 days starting from the day of surgery 1 hour before bedtime.
  The OHRQoL questionnaire comprises 14 questions covering problems the patient may in three main categories: oral function, daily activity, and post-operative symptoms derived from Chaushu's study (Chaushu, Becker, Zeltser, Vasker, & Chaushu, 2004). Patients answered this questionnaire using a 5-category Likert scale (Not at all, Very little, A little, Quite a lot, Very much).

SECONDARY OUTCOMES:
The Modified Dental Anxiety Score (MDAS) | 1 day (Patients completed the modified MDAS once, while waiting for the surgery in the waiting room.)
  The MDAS was used to measure patient anxiety toward dental treatment (Humphris, Dyer, & Robinson, 2009). The MDAS consists of five questions answered with a 5-category Likert scale, ranging from 'not anxious' to 'extremely anxious'. The original MDAS questionnaire does not cover anxiety toward implant surgery. Therefore, a question enquiring about patients' feelings towards implant surgery was added.

CONTACTS AND LOCATIONS:
Overall Officials: Chatchai Kunavisarut, DDS, Study Chair — Department of Advanced General Dentistry, Faculty of Dentistry
Locations (1):
- Faculty of Dentistry, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439
- [Background] Bielemann AM, Marcello-Machado RM, Del Bel Cury AA, Faot F. Systematic review of wound healing biomarkers in peri-implant crevicular fluid during osseointegration. Arch Oral Biol. 2018 May;89:107-128. doi: 10.1016/j.archoralbio.2018.02.013. Epub 2018 Feb 22. PMID 29510331
- [Background] Buser D, Chappuis V, Kuchler U, Bornstein MM, Wittneben JG, Buser R, Cavusoglu Y, Belser UC. Long-term stability of early implant placement with contour augmentation. J Dent Res. 2013 Dec;92(12 Suppl):176S-82S. doi: 10.1177/0022034513504949. Epub 2013 Oct 24. PMID 24158332
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Calvert M, Brundage M, Jacobsen PB, Schunemann HJ, Efficace F. The CONSORT Patient-Reported Outcome (PRO) extension: implications for clinical trials and practice. Health Qual Life Outcomes. 2013 Oct 29;11:184. doi: 10.1186/1477-7525-11-184. PMID 24168680
- [Background] Coolidge T, Hillstead MB, Farjo N, Weinstein P, Coldwell SE. Additional psychometric data for the Spanish Modified Dental Anxiety Scale, and psychometric data for a Spanish version of the Revised Dental Beliefs Survey. BMC Oral Health. 2010 May 13;10:12. doi: 10.1186/1472-6831-10-12. PMID 20465835
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] De Bruyn H, Raes S, Matthys C, Cosyn J. The current use of patient-centered/reported outcomes in implant dentistry: a systematic review. Clin Oral Implants Res. 2015 Sep;26 Suppl 11:45-56. doi: 10.1111/clr.12634. PMID 26385620
- [Background] Feine J, Abou-Ayash S, Al Mardini M, de Santana RB, Bjelke-Holtermann T, Bornstein MM, Braegger U, Cao O, Cordaro L, Eycken D, Fillion M, Gebran G, Huynh-Ba G, Joda T, Levine R, Mattheos N, Oates TW, Abd-Ul-Salam H, Santosa R, Shahdad S, Storelli S, Sykaras N, Trevino Santos A, Stephanie Webersberger U, Williams MAH, Wilson TG Jr, Wismeijer D, Wittneben JG, Yao CJ, Zubiria JPV. Group 3 ITI Consensus Report: Patient-reported outcome measures associated with implant dentistry. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:270-275. doi: 10.1111/clr.13299. PMID 30328187
- [Background] Fortin T, Bosson JL, Isidori M, Blanchet E. Effect of flapless surgery on pain experienced in implant placement using an image-guided system. Int J Oral Maxillofac Implants. 2006 Mar-Apr;21(2):298-304. PMID 16634502
- [Background] Giri J, Pokharel PR, Gyawali R, Bhattarai B. Translation and Validation of Modified Dental Anxiety Scale: The Nepali Version. Int Sch Res Notices. 2017 Jan 29;2017:5495643. doi: 10.1155/2017/5495643. eCollection 2017. PMID 28251175
- [Background] Humphris G, King K. The prevalence of dental anxiety across previous distressing experiences. J Anxiety Disord. 2011 Mar;25(2):232-6. doi: 10.1016/j.janxdis.2010.09.007. Epub 2010 Sep 19. PMID 20952156
- [Background] Humphris GM, Morrison T, Lindsay SJ. The Modified Dental Anxiety Scale: validation and United Kingdom norms. Community Dent Health. 1995 Sep;12(3):143-50. PMID 7584581
- [Background] Iqbal MK, Kim S. A review of factors influencing treatment planning decisions of single-tooth implants versus preserving natural teeth with nonsurgical endodontic therapy. J Endod. 2008 May;34(5):519-29. doi: 10.1016/j.joen.2008.01.002. PMID 18436028
- [Background] Joda T, Derksen W, Wittneben JG, Kuehl S. Static computer-aided implant surgery (s-CAIS) analysing patient-reported outcome measures (PROMs), economics and surgical complications: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:359-373. doi: 10.1111/clr.13136. PMID 30328203
- [Background] McGrath C, Lam O, Lang N. An evidence-based review of patient-reported outcome measures in dental implant research among dentate subjects. J Clin Periodontol. 2012 Feb;39 Suppl 12:193-201. doi: 10.1111/j.1600-051X.2011.01841.x. PMID 22533956
- [Background] Nkenke E, Eitner S, Radespiel-Troger M, Vairaktaris E, Neukam FW, Fenner M. Patient-centred outcomes comparing transmucosal implant placement with an open approach in the maxilla: a prospective, non-randomized pilot study. Clin Oral Implants Res. 2007 Apr;18(2):197-203. doi: 10.1111/j.1600-0501.2006.01335.x. PMID 17348884
- [Background] Sancho-Puchades M, Alfaro FH, Naenni N, Jung R, Hammerle C, Schneider D. A Randomized Controlled Clinical Trial Comparing Conventional And Computer-Assisted Implant Planning and Placement in Partially Edentulous Patients. Part 2: Patient Related Outcome Measures. Int J Periodontics Restorative Dent. 2019 Jul/Aug;39(4):e99-e110. doi: 10.11607/prd.4145. PMID 31226187
- [Background] Sculean A, Gruber R, Bosshardt DD. Soft tissue wound healing around teeth and dental implants. J Clin Periodontol. 2014 Apr;41 Suppl 15:S6-22. doi: 10.1111/jcpe.12206. PMID 24641001
- [Background] Tarnow DP, Cho SC, Wallace SS. The effect of inter-implant distance on the height of inter-implant bone crest. J Periodontol. 2000 Apr;71(4):546-9. doi: 10.1902/jop.2000.71.4.546. PMID 10807116
- [Background] Vercruyssen M, Fortin T, Widmann G, Jacobs R, Quirynen M. Different techniques of static/dynamic guided implant surgery: modalities and indications. Periodontol 2000. 2014 Oct;66(1):214-27. doi: 10.1111/prd.12056. PMID 25123770
- [Background] Vercruyssen M, van de Wiele G, Teughels W, Naert I, Jacobs R, Quirynen M. Implant- and patient-centred outcomes of guided surgery, a 1-year follow-up: An RCT comparing guided surgery with conventional implant placement. J Clin Periodontol. 2014 Dec;41(12):1154-60. doi: 10.1111/jcpe.12305. Epub 2014 Oct 11. PMID 25197015
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Ann Intern Med. 2007 Oct 16;147(8):573-7. doi: 10.7326/0003-4819-147-8-200710160-00010. PMID 17938396
- [Background] Wismeijer D, Joda T, Flugge T, Fokas G, Tahmaseb A, Bechelli D, Bohner L, Bornstein M, Burgoyne A, Caram S, Carmichael R, Chen CY, Coucke W, Derksen W, Donos N, El Kholy K, Evans C, Fehmer V, Fickl S, Fragola G, Gimenez Gonzales B, Gholami H, Hashim D, Hui Y, Kokat A, Vazouras K, Kuhl S, Lanis A, Leesungbok R, van der Meer J, Liu Z, Sato T, De Souza A, Scarfe WC, Tosta M, van Zyl P, Vach K, Vaughn V, Vucetic M, Wang P, Wen B, Wu V. Group 5 ITI Consensus Report: Digital technologies. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:436-442. doi: 10.1111/clr.13309. PMID 30328201
- [Background] Yuan S, Freeman R, Lahti S, Lloyd-Williams F, Humphris G. Some psychometric properties of the Chinese version of the Modified Dental Anxiety Scale with cross validation. Health Qual Life Outcomes. 2008 Mar 25;6:22. doi: 10.1186/1477-7525-6-22. PMID 18364045
- [Result] Chaushu S, Becker A, Zeltser R, Vasker N, Chaushu G. Patients' perceptions of recovery after surgical exposure of impacted maxillary teeth treated with an open-eruption surgical-orthodontic technique. Eur J Orthod. 2004 Dec;26(6):591-6. doi: 10.1093/ejo/26.6.591. PMID 15650068
- [Result] Humphris GM, Dyer TA, Robinson PG. The modified dental anxiety scale: UK general public population norms in 2008 with further psychometrics and effects of age. BMC Oral Health. 2009 Aug 26;9:20. doi: 10.1186/1472-6831-9-20. PMID 19709436